CLINICAL TRIAL: NCT05246059
Title: SARS-CoV-2 Infection/Covid-19 and Anosmia - Prevalence Study, Molecular Analysis and Clinical Trial
Brief Title: Anosmia and Covid-19
Acronym: COVANOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDGE132692; IRAS No. 283758 (Other: NHS Health Research Authority)
Record Dates: First submitted 2022-02-17; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Anosmia; SARS CoV 2 Infection
MeSH Terms: conditions — Anosmia; COVID-19 | interventions — Olfactory Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): 12 weeks of observation, safety information provided
- Treatment (Experimental): 12-weeks of daily olfactory training
  Interventions: Other: Olfactory Training

INTERVENTIONS:
Other: Olfactory Training — Sniffin' Sticks (Duft-Quartett, Burghart Messtechnik, GmbH, Germany)
  Arms: Treatment

SUMMARY:
Our study aims to determine the prevalence of anosmia in patients SARS-Cov-2/Covid-19 infection (both by symptom reporting and smell testing), the efficacy of early olfactory training for the treatment of anosmia caused by infection and the long-term impact of smell dysfunction with a one-year follow-up.

DETAILED DESCRIPTION:
Around 10-15% of patients with acquired anosmia have Post Viral Olfactory Loss (PVOL). Coronaviruses are a known cause for anosmia. At the onset of the COVID-19 pandemic, reports from China, South Korea, US and Europe suggest that a significant proportion of COVID-19 patients describe a loss of smell and taste as the only symptoms or as part of mild flu-like symptoms. It is now well-established that these symptoms are important components of the COVID-19 sequelae with persistent dysfunction described in a subset of individuals.

For this study, individuals, mainly comprising mainly healthcare workers in the UK, with persistent and sudden loss of sense of smell (at least 4 weeks) were recruited to ascertain the prevalence of COVID-19 associated smell dysfunction. A positive COVID-19 test was not a requirement for participation if not readily available nor accessible, however, information regarding COVID-19 antigen and antibody testing was collected post-hoc from those for who data are readily available. All participants (n=227) underwent initial psychophysical smell testing using the Brief Smell Identification Test (BSIT), gustatory testing using Taste Strips and completed the Smell Qx questionnaire. This questionnaire collected relevant demographic information, medical history, details of COVID-19 symptoms experienced, as well as information on olfactory and gustatory function, including those related to quality-of-life.

Participants, who scored 8 or below on the BSIT (indicative of semi-quantitative smell loss) were further invited to participate in the early olfactory training randomized controlled trial. Participants were randomized to undergo either 12 weeks of olfactory training or receive safety information. At the end of the 12-weeks, participants completed a follow-up BSIT and survey.

All participants enrolled at baseline within the eligible timeframe, for whom a valid email address was available, were further invited to participate in 1 year follow-up assessments. This included all participants irrespective of baseline BSIT result and RCT participation. The follow-up included a final electronic survey and BSIT. In addition to questions related to their sense of smell, which were identical to those in the baseline and 12-week follow-up surveys, participants were also asked about any symptoms of long-Covid.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed (positive laboratory antigen test) or suspected COVID-19 infection
* Sudden onset of smell loss
* Smell loss of at least 4 weeks
* Reduced smell function through psycho-physical testing (Brief Smell Identification Test score of 8 or less)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-08-08 (Actual)

PRIMARY OUTCOMES:
Brief Smell Identification Test (BSIT) | 12-weeks
  The absolute difference between the intervention and control arms in BSIT score smell improvement, measured as a change from baseline at 12-weeks.

SECONDARY OUTCOMES:
Quality of Life Score | 12-weeks
  Within subject changes to scoring of questionnaire quality of life items at 12-weeks compared to baseline
Compliance (anecdotal) | 12-weeks
  Participant compliance to olfactory training through anecdotal reporting
Safety (anecdotal) | 12-weeks
  Safety of the use of Sniffin' Sticks through anecdotal reporting

CONTACTS AND LOCATIONS:
Overall Officials: Valerie J. Lund, MD FRCS, Principal Investigator — University College, London; Matt Lechner, MD FRCS, Principal Investigator — University College London, Barts Health NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Barts Health NHS Foundation Trust, London, England
  - Guy's and St. Thomas' NHS Foundation Trust, London, England
  - Wrightington, Wigan and Leigh NHS Foundation Trust, Wigan, England
  - James Paget and Norfolk & Norwich University Hospitals, Gorleston-on-Sea, Great Yarmouth

IPD SHARING:
Plan to Share IPD: No